CLINICAL TRIAL: NCT04839523
Title: An Open, Non-comparative, Multi-center Investigation to Evaluate Performance and Safety of Exufiber Ag+ and Exufiber on Partial Thickness Burns
Brief Title: Performance and Safety of Exufiber Ag+ and Exufiber on Partial Thickness Burns
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTB01
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Partial-thickness Burn

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Wound size and tissue type will be assessed by a single, blinded, third-party clinician. The clinician will use imaging software to measure the size of the wound and identify tissue types, from baseline to last clinical follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Exufiber (Experimental): Treatment with Exufiber gelling fiber dressing
  Interventions: Device: Exufiber
- Exufiber Ag+ (Experimental): Treatment with Exufiber Ag+ silver-coated, gelling fiber dressing
  Interventions: Device: Exufiber Ag+

INTERVENTIONS:
Device: Exufiber — A sterile nonwoven wound dressing made from highly absorbent PVA fibers.
  Arms: Exufiber
Device: Exufiber Ag+ — A sterile nonwoven wound dressing made from highly absorbent PVA fibers, and coated with silver sulphate.
  Arms: Exufiber Ag+

SUMMARY:
This a multi-center, open label, non-comparative, study that will evaluate the clinical safety and performance of Exufiber Ag+ and Exufiber dressings, separately, when used as intended in moderate to high exuding partial thickness burns (PTBs) through assessment of wound progression from baseline to the Subject's last clinical follow-up visit.

Sixty-eight (68) eligible subjects, with moderate to high exuding partial-thickness burns, will be selected for treatment with either Exufiber Ag+ silver-coated gelling dressing, or Exufiber gelling dressing. The study will last 5 weeks, with a requirement of 5 study visits in total, including dressing changes at each study visit.

DETAILED DESCRIPTION:
This is a multi-center study taking place in the United States, and conducted at 3-4 sites/locations. It is designed as an open, non-comparative study to test the safety and performance of Exufiber Ag+ and Exufiber in managing burn healing.

The primary objective of this study is to evaluate the clinical safety and performance of all study dressings, separately, when used as intended in moderate to high exuding partial thickness burns (PTBs) through assessment of wound progression from baseline to the Subject's last clinical follow-up visit. The dressings are intended to promote healing through the management of the wound environment.

Sixty-eight (68) subjects with partial thickness burns will be treated with either Exufiber Ag+ (34 subjects) or Exufiber (34 subjects) primary dressings, at the discretion of the Investigator. Secondary dressings should be non-adherent, non-antimicrobial dressings (local treatment praxis).

Each Subject will be evaluated at five (5) planned study visits for a maximum total treatment period of up to 21 days, unless the burn heals.

Visit 1 is a baseline visit to enroll Subjects and determine burn extent. Each Subject will be assigned to either Exufiber Ag+ or Exufiber primary dressings and treated according to the Instructions for Use (IFU) and the local clinical routine.

Visit 2 is a Confirmation Visit at up to 3 days, where the Investigator will confirm the burn meets study eligibility, and has not progressed to a full-thickness burn.

Visits 3, 4, and 5 are follow-up visits at days 7, 14, and 21, respectively, from the date of the primary dressing application.

At each follow-up visit the Subject will return to the clinic for evaluation and primary dressing change. Wound progression will be determined by the Investigator at each study visit and measured by three outcome variables (Deteriorated, No Change, Improved). Images of the wound at each follow up visit will be analyzed to determine changes in wound size.

Secondary endpoints will be collected identically at each visit at each clinical site to assess safety and performance of the dressings. The secondary objectives are:

* To evaluate time to discontinuation of study dressings from baseline to the last clinical follow-up visit, up to 21 days.
* To evaluate clinical outcomes of the study wound from baseline to the last clinical visit up to 21 days.
* To evaluate epithelization from baseline to the last clinical follow-up visit up to 21 days based on digital photo imaging software measurements.
* To evaluate a change in wound size from baseline to the last clinical follow-up visit up to 21 days based on digital photo and imaging software measurements.
* To evaluate healing status, including exudate levels, infection status, and proportion of burn healed, by clinician's visual judgement, at Confirmation Visit (up to 72 hours) and at each clinic follow-up visit, up to 21 days.
* To evaluate Subject-reported pain at application, during wear, and at dressing changes through questionnaires at each clinic follow-up visit up to 21 days.
* To evaluate treatment and dressing selections, including type and quantity, at application and at each clinic follow-up visit up to 21 days.
* To evaluate clinician handling of the dressing at application and at every dressing change performed at the clinic, from baseline and at each follow-up visit up to 21 days.
* To evaluate clinician assessment of the dressing at application and at every dressing change performed at the clinic, from baseline and at each follow-up visit up to 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Burn of thermal origin
3. Patients presenting with partial thickness burns covering < 5% TBSA for study treatment
4. TBSA covered with any burn type is ≤15%, with a maximum of 10% being full thickness burns
5. Clean wounds with ≤10% necrotic tissue
6. Patients presenting with moderate to high exuding wounds
7. Serous or Serosanguinous exudate
8. Patient is not contraindicated for the dressing to which he/she is assigned

Exclusion Criteria:

1. Electrical Burns
2. Chemical Burns including acidic or basic sources
3. Ionizing radiation injuries
4. Dry wounds
5. Neonates
6. Patients with delayed presentation for burn care (>72 hours from time of injury)
7. Before entry into the study, treatment to the study wound included an active agent that would confound study results, as determined by the Investigator
8. Burns under study treatment transitioning to full thickness, or deep partial thickness burns requiring surgical treatment
9. Clinically infected burn
10. Patients with insulin dependent diabetes mellitus
11. Patients treated with systemic glucocorticosteroids, except patients taking occasional doses or doses less than 10mg prednisolone per day or equivalent
12. Patients who have used immunosuppressive agents, radiation or chemotherapy within past 30 days
13. Known allergy/hypersensitivity to any of the components of the investigation products
14. History of comorbid conditions or diagnoses associated with higher risk of infection as determined by the Investigator
15. Diagnosed underlying disease(s) (e.g. HIV/AIDS, cancer, severe anemia)
16. Patients that are not expected to comply with the investigation due to physical and/or mental conditions
17. Pregnancy
18. Participation in other clinical investigation(s) within 1 month prior to start of the investigation
19. Previously enrolled in this investigation

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound progression | 5 weeks
  A subjective measurement to determine wound progression since the last visit, determined by three outcome variables:
  Deteriorated
  No Change
  Improved

SECONDARY OUTCOMES:
Time to discontinuation of study dressings | 5 weeks
  Measured by time (in days) from baseline to last clinical follow-up
Wound Size | 5 weeks
  Wound size (measured in inches or centimeters), at each study visit, from baseline to last clinical follow-up, using planimetry software to obtain measurements from digital photographs. Measurements to include length, width, and depth.
Re-epithelialization of wound | 5 weeks
  A measure of re-epithelization tissue, as a percentage of wound, from baseline to last clinical follow-up, using planimetry software to obtain measurements from digital photographs.
Wound Exudate | 5 weeks
  Evaluate the level of wound exudate, using the variables listed below:
  Dry
  Moist
  Wet
  Saturated
  Leaking
Wound Maceration | 5 weeks
  Determine the presence of wound maceration, using the variables listed below:
  Yes
  No
Proportion of Burn Healed | 5 weeks
  Evaluate the proportion of the burn that is healed, by clinician judgement, using the variables listed below:
  No healing
  0-30% healed
  31-70% healed
  71-99% healed
  100% healed
Blistering | 5 weeks
  Determine the presence of wound blistering, using the variables listed below:
  Yes
  No
Wound Redness/Irritation peri-wound skin | 5 weeks
  Determine the presence of redness and irritation on the peri-wound skin, using the variables listed below:
  Yes
  No
Exudate Nature | 5 weeks
  Determine the nature of wound exudate, using the variables listed below:
  Serous
  Serosanguinous
  Sanguineous
  Purulent
Malodor | 5 weeks
  Determine the presence of wound malodor, using the variables listed below:
  None
  Slight
  Moderate
  Strong
Burn odor | 5 weeks
  Determine the presence of burn odor, using the variables listed below:
  Yes
  No
Local infection | 5 weeks
  Determine the presence of signs of local wound infection, using the variables listed below:
  New / Increasing Pain
  Delayed / Stalled Healing
  Purulent discharge
  Erythema
  Local Warmth
  Exudation
  Odor
  Pyrexia
  Induration
  Leukocytosis
  Edema / Swelling
  Eschar
Subject pain | 5 weeks
  Measured at dressing application, change, and removal, using a patient reported outcome questionnaire that is used to evaluate pain intensity on a validated scale from 0-10. A higher score correlates with greater experienced pain.
Dressing Adherence | 5 weeks
  Subjective measurement to asses performance of the primary dressing and its adherence to the wound bed, using the variables listed below:
  Yes
  No
Rewetting | 5 weeks
  Subjective measurement to asses performance of the primary dressing and the need for re-wetting prior to removal, using the variables listed below:
  Yes
  No
Dressing ability to rehydrate | 5 weeks
  Subjective measurement to asses performance of the primary dressing and its ability to rehydrate the wound, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing ability to retain exudate | 5 weeks
  Subjective measurement to asses performance of the primary dressing and its ability to retain wound exudate, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing ability to absorb blood | 5 weeks
  Subjective measurement to asses performance of the primary dressing and its ability to absorb blood, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing ability to retain slough | 5 weeks
  Subjective measurement to asses performance of the primary dressing and its ability to retain slough, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing ability to clean wound bed | 5 weeks
  Subjective measurement to asses performance of the primary dressing and its ability to clean the wound bed, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing ability to retain gelling properties | 5 weeks
  Subjective measurement to asses performance of the primary dressing and its ability to retain its gelling properties, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing ability to retain balanced moist environment | 5 weeks
  Subjective measurement to asses performance of the primary dressing and its ability to retain a balanced moist environment, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing conformability | 5 weeks
  Subjective measurement to assess performance of the primary dressing and its ability to conform, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing flexibility | 5 weeks
  Subjective measurements to assess performance of the primary dressing and its flexibility, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Ease of dressing application | 5 weeks
  Subjective measurement to assess the handling of the primary dressing and ease of dressing application, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Ease of dressing removal with and without moistening | 5 weeks
  Subjective measurement to assess the handling of the primary dressing and ease of removal with and without moistening, using the variables listed below:
  Very poor
  Poor
  Good
  Very good
  N/A
Dressing removal in one piece | 5 weeks
  Subjective measurement to assess the handling of primary dressing and its ability to be removed in one piece, using the variables listed below:
  Yes
  No
Residuals of dressing material in the wound or surrounding skin | 5 weeks
  Subjective measurement to assess presence of primary dressing residuals in the wound or surrounding skin at the time of removal, using the variables listed below:
  Yes
  No
Bleeding at removal | 5 weeks
  Subjective measurement to assess presence of bleeding at the time of primary dressing removal, using the variables listed below:
  Yes
  No

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Arizona Burn Center, Valleywise Health, Phoenix, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - University of South Florida-Tampa General Hospital, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Drexel Univerisity, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No